CLINICAL TRIAL: NCT05535231
Title: A Randomized, Double-Blinded, Comparator-Controlled, Crossover Study to Evaluate the Pharmacokinetics of Gaia Full-Spectrum Turmeric Phytocapsules
Brief Title: A Study to Evaluate the Effect of Turmeric in Healthy Participants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gaia Herbs Inc. (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: G02-21-01-T0030
Record Dates: First submitted 2022-09-06; First posted 2022-09-10 (Actual); Last update posted 2023-02-24 (Actual); Status verified 2023-02

CONDITIONS: Healthy
Keywords: Turmeric; Curcumin

STUDY DESIGN:
Intervention Model Description: Randomization at 1:1 ratio for test product or comparator
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Turmeric test product (Experimental): Turmeric
  Interventions: Dietary Supplement: Turmeric test product
- Turmeric comparator (Active Comparator): Turmeric
  Interventions: Dietary Supplement: Turmeric comparator

INTERVENTIONS:
Dietary Supplement: Turmeric test product — 2 capsules of 490 mg Turmeric are taken with water once
  Other Names: Turmeric Supreme Extra Strength
  Arms: Turmeric test product
Dietary Supplement: Turmeric comparator — 2 capsules of 200 mg Turmeric are taken with water once
  Other Names: Renew Actives Turmeric Curcumin
  Arms: Turmeric comparator

SUMMARY:
Turmeric is recognized as a bioactive compound with potential benefits for human health. This study compares the pharmacokinetic profile of the Turmeric test product to a comparator.

DETAILED DESCRIPTION:
This randomized, double-blinded, comparator-controlled, crossover study will compare the pharmacokinetic profile of the Turmeric test product to a comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult participants who are 18 to 49 years of age (inclusive).
2. In good general health (no active or uncontrolled diseases or conditions) and is able to consume the study product.
3. Have a body mass index between 18.5 to 24.9 kg/m2 (inclusive).
4. Have normal or acceptable to the investigator heart rate at screening.
5. Individuals with childbearing potential should have a negative pregnancy test at baseline and must agree to practice an acceptable form of non-hormonal birth control throughout the study, including but not limited to:

   1. double-barrier method
   2. non-hormonal intrauterine devices
   3. complete abstinence from sexual intercourse that can result in pregnancy
   4. vasectomy of partner at least 6 months prior to the first dose of study product Individuals with the potential to impregnate others must agree to use condoms or other acceptable methods to prevent pregnancy throughout the study. Complete abstinence from sexual intercourse that can result in pregnancy is also acceptable.
6. Must have suitable veins for repeated venipuncture.
7. Able to swallow pills or capsules whole and without chewing.
8. Willing and able to comply with the protocol, including:

   * Agrees to consume the standardized meals provided at the site during Visit 2 and Visit 3
   * Agrees to fast overnight, i.e., no food or liquids for a minimum of 10 hours prior to dosing (except for water, permitted up to 1-hour prior to dosing) on Visit 2 and Visit 3
   * Agrees to refrain from consuming grapefruit, pomelo, Seville orange, and starfruit containing foods/beverages 7 days prior to Visit 2 and throughout the study
   * Agrees to refrain from caffeine/xanthine and alcohol or alcohol-containing products 48 hours prior to dosing on Visit 2 and Visit 3
   * Agrees to refrain from the use/application of treatments/procedures listed in the protocol
   * Agrees to maintain the same diet and exercise habits throughout the study
   * Agrees not to donate blood or plasma for 30 days after completing the study
   * Able to give voluntary consent

Exclusion Criteria:

1. Participants who are lactating, pregnant or planning to become pregnant during the study.
2. Have a known sensitivity, intolerability, or allergy to any of the standardized study meals/snacks, study products or their excipients.
3. Received a vaccine for COVID-19 in the 2 weeks prior to screening or during the study period, current COVID-19 infections, or currently have the post COVID-19 condition as defined by World Health Organization (i.e., individuals with a history of probable or confirmed SARS-CoV-2 infection, usually 3 months from the onset of COVID-19 with symptoms that last for at least 2 months and cannot be explained by an alternative diagnosis). Note: screened participants who have received a COVID-19 vaccine 2 weeks prior to screening would be eligible to participate after completing a 14-day washout period.
4. Have uncontrolled or controlled high blood pressure (≥140 systolic or ≥90 diastolic mmHg) at screening.
5. Have a history of heart disease/cardiovascular disease, renal or hepatic impairment/disease, diabetes (Type I or Type II), previously diagnosed or current diagnosis of any psychiatric disorders, unstable thyroid disease, immune disorders and/or immunocompromised (e.g. HIV/AIDS), cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to the screening visit, or any clinically significant disease or disorder which, in the opinion of the investigator, may either put the potential participant at risk because of participation in the study, or influences the results or the potential participant's ability to participate in the study.
6. Major surgery with general anesthesia in the 3 months prior to screening or planned major surgery during the course of the study.
7. Have a history of blood clotting disorders.
8. Reports a significant blood loss or blood donation totaling between 101 mL to 449 mL of blood within 30 days prior to the first pharmacokinetic visit or a blood donation of more than 450 mL within 56 days prior to the first pharmacokinetic visit.
9. Reports donating plasma (e.g., plasmapheresis) within 15 days prior to the first pharmacokinetic visit.
10. Have an abnormality or obstruction of the gastrointestinal tract precluding swallowing (e.g., dysphagia) and digestion (e.g., known intestinal malabsorption, celiac disease, inflammatory bowel disease, chronic pancreatitis, steatorrhea).
11. Have gallstones, bile duct obstruction, stomach ulcers, excess stomach acid, or gastroesophageal reflux disease.
12. History of alcohol or substance abuse in the 12 months prior to screening or use that to the opinion of the Qualified Investigator may be of a concern for the study.
13. Receipt or use of test product(s) in another research study within 28 days prior to baseline or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
14. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2022-09-24 (Actual); Primary Completion 2022-10-03 (Actual); Study Completion 2022-10-03 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics- Area under the plasma concentration-time curve for 8 hours (AUC0-8h) | 8 hours
  Test products area under the plasma concentration-time curve for 8 hours (AUC0-8h)
Pharmacokinetics- Peak plasma concentration (Cmax) | 8 hours
  Test products Peak plasma concentration (Cmax)
Pharmacokinetics- Time to reach Cmax (Tmax) | 8 hours
  Test products Time to reach Cmax (Tmax)

SECONDARY OUTCOMES:
Pharmacokinetics- Total area under the curve (observed from 0-8 hours, and extrapolated from 8 hours to infinity) [AUC(0-∞)] | 8 hours
  Test products Total area under the curve (observed from 0-8 hours, and extrapolated from 8 hours to infinity) [AUC(0-∞)]
Pharmacokinetics- Half-life (T1/2) | 8 hours
  Test products Half-life (T1/2)
Pharmacokinetics- Terminal elimination rate constant (Kel) | 8 hours
  Test products Terminal elimination rate constant (Kel)
Safety- participants experiencing adverse events | 8 days
  The number of participants experiencing Treatment Emergent Adverse Events (TEAEs)
Safety- adverse events | 8 days
  The total number Treatment Emergent Adverse Events (TEAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Bier, MD, Principal Investigator — Nutrasource Pharmaceutical and Nutraceutical Services, Inc.
Locations (1):
- Nutrasource Clinical Trial Site, Guelph, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No